CLINICAL TRIAL: NCT00649506
Title: Single-Dose Food In Relative Bioavailability Study of Mylan Nitrofurantoin Macrocrystals 100 mg Capsules and Procter & Gamble Macrodantin® 100 mg Capsules in Healthy Volunteers
Brief Title: Food Study of Nitrofurantoin Macrocrystals 100 mg Capsules and Macrodantin® 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullvan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NITF-0324
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Nitrofurantoin

ARMS (2):
- 1 (Experimental): Nitrofurantoin Macrocrystals 100 mg Capsules
  Interventions: Drug: Nitrofurantoin Macrocrystals 100 mg Capsules
- 2 (Active Comparator): Macrodantin® 100 mg Capsules
  Interventions: Drug: Macrodantin® 100 mg Capsules

INTERVENTIONS:
Drug: Nitrofurantoin Macrocrystals 100 mg Capsules — 100mg, single dose fed
  Arms: 1
Drug: Macrodantin® 100 mg Capsules — 100mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to evaluate the relative bioavailability of Mylan's nitrofurantoin macrocrystals 100 mg capsules to Procter & Gamble's Macrodantin® 100 mg capsules following a single, oral 100 mg (1 x 100 mg) dose in 28 healthy, adult, non-tobacco using volunteers under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male and/or non-pregnant, non-lactating female

   1. Women of childbearing potential must have negative serum Beta-human chorionic gonadotropin (HCG) pregnancy tests performed within 14 days prior to of the study and on the evening prior to each dose administration. If dosing is scheduled on Sunday or Monday, the HCG pregnancy test should be given within 48 hours prior to dosing of each study period. An additional serum (Beta-HCG) pregnancy test will be performed upon completion of the study.
   2. Women of childbearing potential must practice abstinence or be using an acceptable form of contraception throughout the duration of the study. Acceptable forms of contraception include the following:

      1. intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
      2. barrier methods containing or used in conjunction with a spermicidal agent, or
      3. postmenopausal or surgical sterility accompanied with a documented postmenopausal course of at least one year (tubal ligation, oophorectomy or hysterectomy).

      Note: Hormonal contraceptives are NOT an acceptable form of contraception in this study.
   3. During the course of the study, from study screen until study exit - including the washout period, women of childbearing potential must use a spermicide containing barrier method of contraception in addition to their current contraceptive method. This advice should be documented in the informed consent form.
3. Weight: At least 60 kg (132 lbs) for man and 48 kg (106 lbs) for women and within 15% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, 12-lead ECG, hepatitis B and hepatitis C tests, HIV test, and urine drug screen including amphetamine, barbiturates, benzodiazepine, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the initial dose of study medication.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within the 48 hours prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
3. Medications:

   1. Use of any medication within the 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 30 days of the initial dose of study medication.
   3. Use of hormonal contraceptives or hormonal replacement therapy within 3 months of the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease.
   2. History of drug and/or alcohol abuse.
   3. Acute illness at the time of either the pre-study medical evaluation or dosing.
   4. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to nitrofurantoin or other related products.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Use of antacids containing magnesium trisilicate within 2 days of dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Clark, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html